CLINICAL TRIAL: NCT04240041
Title: Accuracy of Trans-cerebellar Diameter and Placental Thickness in Third Trimesteric Pregnant Women for Calculation of Gestational Age: Prospective Study
Brief Title: Trans-cerebellar Diameter and Placental Thickness in Third Trimesteric Pregnant Women for Calculation of Gestational Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayatullah Abd ElFatah Mahmoud, Resident of O&G, Ain Shams University
Other Study IDs: TCD/PT-GA
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Gestational Age and Weight Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women at 32-36 weeks gestational age: Pregnant women at 32-36 weeks gestational age with sure dates and crown-rump length dating ultrasound
  Interventions: Diagnostic Test: Transcerebellar diamater; Diagnostic Test: Placental thickness

INTERVENTIONS:
Diagnostic Test: Transcerebellar diamater — Using SAMSUNG H60 convex probe 2-8 MHz Machine by the same sonographer, trans-cerebellar diameter is identified by obtaining an oblique view through posterior fossa that included visualization of midline thalamus, cerebellar hemispheres and cisterna magna.
Diagnostic Test: Placental thickness — Using SAMSUNG H60 convex probe 2-8 MHz Machine by the same sonographer, placental thickness will be measured at the level of the umbilical cord insertion excluding the myometrium and sub-placental veins

SUMMARY:
Pregnant women at 32-36 weeks gestational age with sure gestational dating (based in both last menstrual period and dating ultrasound) and otherwise normal singleton pregnancy will be recruited. Ultrasonographic estimation of gestational age using combined transcerebellar diameter and placental thickness will be compared to the actual estimated gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Sure of dates
* Have dating ultrasound with crown rump length between (9 to 12 )weeks
* No hormonal contraception 3 months before conception.
* Regular menstrual cycles.
* Medically free.
* Single pregnancy
* Gestational age 32-36 weeks

Exclusion Criteria:

* Irregular menstrual cycles and not sure of dates
* Multiple pregnancy.
* Fetal anomalies.
* Placenta previa, placental anomalies and poor visualization of the placenta
* Fetal growth restriction
* Pregnant women with medical disorder e.g. diabetes mellitus, Pre-eclampsia, Systemic lupus erythromatosis, hypertension.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women at 32-36 weeks gestational age with sure gestational dating (based in both last menstrual period and dating ultrasound) and otherwise normal singleton pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Concordance between estimated gestational age and combined transcerebellar diameter and placental thickness estimation | 32-36 weeks gestational age
  Concordance between the estimated gestational age using last menstrual period and dating ultrasound; and that estimated using combination of transcerebellar diameter and placental thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ayat Allah Mahmoud, MB BCh, Principal Investigator — Resident of Obstetrics & Gynecology
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Abbsia, Egypt

IPD SHARING:
Plan to Share IPD: No